CLINICAL TRIAL: NCT03117543
Title: Screening and Diagnostic Approaches in Gestational Diabetes (GDM) and the Impact of Ethnicity on Markers of Glycaemia in Pregnancy
Brief Title: Diagnostic Approaches in Gestational Diabetes and Impact of Ethnicity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other); Collaboration for Leadership in Applied Health Research and Care, United Kingdom (Unknown)
Responsible Party: Sponsor
Other Study IDs: KCH16-035; 15/LO/1494 (Other: Health Research Authority Research Ethics Committee); 180588 (Other: IRAS)
Record Dates: First submitted 2016-07-11; First posted 2017-04-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Diabetes, Gestational
Keywords: Screening
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples, fasting and at 60 min and 120 min post 75g oral glucose.
Oversight: Data Monitoring Committee: No

SUMMARY:
Gestational diabetes (GDM) means raised blood glucose found for the first time in pregnancy. GDM is common, particularly in women from minority ethnicities. GDM does not cause any symptoms in the mother. GDM is associated with adverse pregnancy outcomes which can be improved with treatment of GDM. The United Kingdom National Institute for Health and Care Excellence (NICE) recommend pregnant women with one or more risk factors should have a 75g oral glucose tolerance test (OGTT). The OGTT is performed in a clinic with venous plasma glucose measured fasting and at 2 hours. This is resource-intensive, and some women with GDM may be missed by this risk-factor based approach. The International Association of Diabetes and Pregnancy Study Groups (IADPSG 2010) recommends screening all pregnant women with 2-hour, 3 sample (fasting, 1 and 2 hour), 75g OGTT, which is even more resource intensive. Developing more cost-effective and convenient approaches to screening for GDM is a priority.

The researchers will validate a new home-use OGTT system (hOGTT), which measures whole blood glucose in capillary blood ('finger-stick' sample), against the gold standard venous plasma glucose in pregnancy.

The researchers will also investigate the performance of glycated haemoglobin (HbA1c) in screening for GDM. HbA1c is used for diagnosis of diabetes outside of pregnancy, but is currently not recommended for screening for GDM.

The researchers will also investigate relationships between glucose measured in different samples (venous versus capillary), different fractions (plasma versus whole blood), and using different methods in pregnancy.

In a substudy the researchers will investigate: ethnic differences in HbA1c and other glycaemic markers; the contribution of fasting and postprandial glucose handling, diet and ethnicity on HbA1c; and ethnic differences in insulin responses to 75g OGTT in pregnancy.

The researchers will invite pregnant women between 16-34 weeks gestation to participate. The research involves one hospital visit for an OGTT. Participants will have venous blood samples taken fasting and at 1-hour and 2-hours, and at the same times finger-stick blood samples will be tested. The researchers will invite women of Black African, Black Caribbean and White European ethnicity to participate in a substudy in which participants will have extra blood taken and a diet assessment.

If the hOGTT provides accurate results in pregnancy, using it to perform OGTTs at home would make screening for GDM less expensive and more convenient and may facilitate universal screening for GDM. Understanding ethnic differences in HbA1c will help determine if HbA1c is a reliable screening tool for GDM in our ethnically diverse local population.

ELIGIBILITY:
Inclusion Criteria:

Main study:

* Pregnant woman at least 18 years of age
* 16-34 weeks gestation.
* Booked for pregnancy care at a participating centre
* Able to give informed consent to participate

Substudy:

In addition to the inclusion criteria of main study:

• Women who are of White European, Black African or Black Caribbean ethnicity.

Exclusion Criteria:

Main study

* Unable to give informed consent
* Known pre-pregnancy diabetes
* GDM diagnosed in the current pregnancy

Substudy

In addition to main study criteria:

* Women known to have sickle cell anaemia or thalassaemia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of hOGTT venous plasma equivalent glucose (hOGTT-VPEqG) results within ±10% of paired venous plasma glucose measured on a YSI analyser (VPG-YSI) (reference standard). | Each participant is studied on one occasion between 16-34 weeks gestation.
  hOGTT-VPEqG (in mmol/l) is capillary whole blood glucose measured on the home Oral Glucose Tolerance Test (hOGTT) system (the device being evaluated) expressed as venous plasma equivalent glucose (VPEqG).
  VPG-YSI (in mmol/l) is venous plasma glucose measured on YSI 2300 Stat Analyser (YSI Life Sciences), a recognised reference standard, average of 2 measurements.
  Paired means samples taken at the same time.
  Results will be reported for glucose (VPG-YSI) range 4.5-11mmol/L. This was chosen because it encompasses the GDM diagnostic cut-offs for both National Institute for Health and Care Excellence (NICE) 2015 and International Association of Diabetes and Pregnancy Study Groups (IADPSG) 2010 criteria.
  Samples taken fasting and at 1 hour and 2 hours post 75g oral glucose load will be considered together in this analysis.

SECONDARY OUTCOMES:
Percentage of hOGTT venous plasma equivalent glucose (hOGTT-VPEqG) results within ±15% of paired venous plasma glucose measured on a YSI analyser (VPG-YSI) (reference standard). | Each participant is studied on one occasion between 16-34 weeks gestation.
  hOGTT-VPEqG (in mmol/l) is capillary whole blood glucose measured on the home Oral Glucose Tolerance Test (hOGTT) system (the device being evaluated) expressed as venous plasma equivalent glucose (VPEqG).
  VPG-YSI (in mmol/l) is venous plasma glucose measured on YSI 2300 Stat Analyser (YSI Life Sciences), a recognised reference standard, average of 2 measurements.
  Paired means samples taken at the same time.
  Results will be reported for glucose (VPG-YSI) range 4.5-11mmol/L. This was chosen because it encompasses the GDM diagnostic cut-offs for both National Institute for Health and Care Excellence (NICE) 2015 and International Association of Diabetes and Pregnancy Study Groups (IADPSG) 2010 criteria.
  Samples taken fasting and at 1 hour and 2 hours post 75g oral glucose load will be considered together in this analysis.
Percentage of hOGTT venous plasma equivalent glucose (hOGTT-VPEqG) results within ±20% of paired venous plasma glucose measured on a YSI analyser (VPG-YSI) (reference standard). | Each participant is studied on one occasion between 16-34 weeks gestation.
  hOGTT-VPEqG (in mmol/l) is capillary whole blood glucose measured on the home Oral Glucose Tolerance Test (hOGTT) system (the device being evaluated) expressed as venous plasma equivalent glucose (VPEqG).
  VPG-YSI (in mmol/l) is venous plasma glucose measured on YSI 2300 Stat Analyser (YSI Life Sciences), a recognised reference standard, average of 2 measurements.
  Paired means samples taken at the same time.
  Results will be reported for glucose (VPG-YSI) range 4.5-11mmol/L. This was chosen because it encompasses the GDM diagnostic cut-offs for both National Institute for Health and Care Excellence (NICE) 2015 and International Association of Diabetes and Pregnancy Study Groups (IADPSG) 2010 criteria.
  Samples taken fasting and at 1 hour and 2 hours post 75g oral glucose load will be considered together in this analysis.
Sensitivity of the hOGTT system for diagnosis of GDM using NICE 2015 criteria (gold standard VPG-YSI). | Each participant is studied on one occasion between 16-34 weeks gestation.
  VPG-YSI is venous plasma glucose measured on YSI 2300 Stat Analyser (YSI Life Sciences), a recognised reference standard, average of 2 measurements.
  NICE (National Institute for Health and Care Excellence) 2015 diagnostic criteria for GDM are: fasting venous plasma glucose ≥ 5.6mmol/L, 2-hour post 75g oral glucose venous plasma glucose ≥ 7.8mmol/L.
Specificity of the hOGTT system for diagnosis of GDM using NICE 2015 criteria (gold standard VPG-YSI). | Each participant is studied on one occasion between 16-34 weeks gestation.
  VPG-YSI is venous plasma glucose measured on YSI 2300 Stat Analyser (YSI Life Sciences), a recognised reference standard, average of 2 measurements.
  NICE (National Institute for Health and Care Excellence) 2015 diagnostic criteria for GDM are: fasting venous plasma glucose ≥ 5.6mmol/L, 2-hour post 75g oral glucose venous plasma glucose ≥ 7.8mmol/L.
Sensitivity of the hOGTT system for diagnosis of GDM using IADPSG 2010 criteria (gold standard VPG-YSI). | Each participant is studied on one occasion between 16-34 weeks gestation.
  VPG-YSI is venous plasma glucose measured on YSI 2300 Stat Analyser (YSI Life Sciences), a recognised reference standard, average of 2 measurements.
  IADPSG (the International Association of Diabetes and Pregnancy Study Groups) 2010 diagnostic criteria for GDM are: 1 or more of fasting venous plasma glucose ≥ 5.1mmol/L, 1-hour post 75g oral glucose venous plasma glucose ≥ 10.0mmol/L or 2-hour post 75g oral glucose venous plasma glucose ≥ 8.5mmol/L.
Specificity of the hOGTT system for diagnosis of GDM using IADPSG 2010 criteria (gold standard VPG-YSI). | Each participant is studied on one occasion between 16-34 weeks gestation.
  VPG-YSI is venous plasma glucose measured on YSI 2300 Stat Analyser (YSI Life Sciences), a recognised reference standard, average of 2 measurements.
  IADPSG (the International Association of Diabetes and Pregnancy Study Groups) 2010 diagnostic criteria for GDM are: 1 or more of fasting venous plasma glucose ≥ 5.1mmol/L, 1-hour post 75g oral glucose venous plasma glucose ≥ 10.0mmol/L or 2-hour post 75g oral glucose venous plasma glucose ≥ 8.5mmol/L.
Relationship between whole blood and plasma glucose in capillary blood samples in pregnancy. | Each participant is studied on one occasion between 16-34 weeks gestation.
  In capillary blood samples, glucose will be measured in both whole blood and plasma on the YSI analyser. The relationship between whole blood and plasma glucose measurements will be reported.
Relationship between whole blood and plasma glucose in venous blood samples in pregnancy. | Each participant is studied on one occasion between 16-34 weeks gestation.
  In venous blood samples, glucose will be measured in both whole blood and plasma on the YSI analyser. The relationship between whole blood and plasma glucose measurements will be reported.
Relationship between capillary whole blood and venous whole blood glucose in pregnancy. | Each participant is studied on one occasion between 16-34 weeks gestation.
  Glucose will be measured on the YSI analyser in paired capillary whole blood and venous whole blood samples. The relationship between capillary and venous whole blood glucose will be reported.
  Paired means samples taken at the same time.
Relationship between capillary plasma glucose and venous plasma glucose in pregnancy. | Each participant is studied on one occasion between 16-34 weeks gestation.
  Glucose will be measured on the YSI analyser in paired capillary plasma and venous plasma samples. The relationship between capillary and venous plasma glucose will be reported.
  Paired means samples taken at the same time.
Sensitivity of HbA1c for screening for GDM versus gold standard of 75g OGTT and VPG-YSI measurement (NICE 2015 criteria). | Each participant is studied on one occasion between 16-34 weeks gestation.
  HbA1c (haemoglobin A1c, glycated haemoglobin) measured on venous whole blood in a hospital laboratory (IFCC standardised).
  VPG-YSI is venous plasma glucose measured on YSI 2300 Stat Analyser (YSI Life Sciences), a recognised reference standard, average of 2 measurements.
  NICE (National Institute for Health and Care Excellence) 2015 diagnostic criteria for GDM are: fasting venous plasma glucose ≥ 5.6mmol/L, 2-hour post 75g oral glucose venous plasma glucose ≥ 7.8mmol/L.
Specificity of HbA1c for screening for GDM versus gold standard of 75g OGTT and VPG-YSI measurement (NICE 2015 criteria). | Each participant is studied on one occasion between 16-34 weeks gestation.
  HbA1c (haemoglobin A1c, glycated haemoglobin) measured on venous whole blood in a hospital laboratory (IFCC standardised).
  VPG-YSI is venous plasma glucose measured on YSI 2300 Stat Analyser (YSI Life Sciences), a recognised reference standard, average of 2 measurements.
  NICE (National Institute for Health and Care Excellence) 2015 diagnostic criteria for GDM are: fasting venous plasma glucose ≥ 5.6mmol/L, 2-hour post 75g oral glucose venous plasma glucose ≥ 7.8mmol/L.
Sensitivity of HbA1c for screening for GDM versus gold standard of 75g OGTT and VPG-YSI measurement (IADPSG 2010 criteria). | Each participant is studied on one occasion between 16-34 weeks gestation.
  HbA1c (haemoglobin A1c, glycated haemoglobin) measured on venous whole blood in a hospital laboratory (IFCC standardised).
  VPG-YSI is venous plasma glucose measured on YSI 2300 Stat Analyser (YSI Life Sciences), a recognised reference standard, average of 2 measurements.
  IADPSG (the International Association of Diabetes and Pregnancy Study Groups) 2010 diagnostic criteria for GDM are: 1 or more of fasting venous plasma glucose ≥ 5.1mmol/L, 1-hour post 75g oral glucose venous plasma glucose ≥ 10.0mmol/L or 2-hour post 75g oral glucose venous plasma glucose ≥ 8.5mmol/L.
Specificity of HbA1c for screening for GDM versus gold standard of 75g OGTT and VPG-YSI measurement (IADPSG 2010 criteria). | Each participant is studied on one occasion between 16-34 weeks gestation.
  HbA1c (haemoglobin A1c, glycated haemoglobin) measured on venous whole blood in a hospital laboratory (IFCC standardised).
  VPG-YSI is venous plasma glucose measured on YSI 2300 Stat Analyser (YSI Life Sciences), a recognised reference standard, average of 2 measurements.
  IADPSG (the International Association of Diabetes and Pregnancy Study Groups) 2010 diagnostic criteria for GDM are: 1 or more of fasting venous plasma glucose ≥ 5.1mmol/L, 1-hour post 75g oral glucose venous plasma glucose ≥ 10.0mmol/L or 2-hour post 75g oral glucose venous plasma glucose ≥ 8.5mmol/L.

OTHER OUTCOMES:
HbA1c in pregnant women of Black (Black African and Black Caribbean) compared to White European ethnicity. | Each participant in this sub-study is studied on one occasion between 16-34 weeks gestation.
  HbA1c (haemoglobin A1c, glycated haemoglobin) will be measured on venous whole blood in a hospital laboratory (IFCC standardised).
  Mean HbA1c in pregnant women of Black (Black African and Black Caribbean) and White European ethnicity will be reported and compared using a t test.
Fructosamine in pregnant women of Black (Black African and Black Caribbean) compared to White European ethnicity. | Each participant in this sub-study is studied on one occasion between 16-34 weeks gestation.
  Serum fructosamine will be measured using commercially available assays. Mean fructosamine in pregnant women of Black (Black African and Black Caribbean) and White European ethnicity will be reported and compared using a t test.
The independent factors (out of fasting venous plasma glucose; 1 hour post 75g oral glucose venous plasma glucose; 2 hour post 75g oral glucose venous plasma glucose; dietary carbohydrate content; gestation; or ethnicity) that predict HbA1c in pregnancy. | Each participant in this sub-study is studied on one occasion between 16-34 weeks gestation.
  HbA1c (haemoglobin A1c, glycated haemoglobin) will be measured on venous whole blood in a hospital laboratory (IFCC standardised).
  Multiple regression analysis will be conducted. Independent variables to be included in the model include: fasting venous plasma glucose measured on a YSI analyser; 1 hour post 75g oral glucose venous plasma glucose measured on a YSI analyser; 2 hour post 75g oral glucose venous plasma glucose measured on a YSI analyser; dietary carbohydrate content (measured using a face-to-face structured 48 hour dietary recall interview using the triple pass methodology of the Medical Research Council); gestation; and ethnicity.
Serum insulin concentration at 60 min after 75g oral glucose in pregnant women of Black (Black African and Black Caribbean) compared to White European ethnicity. | Each participant in this substudy is studied on one occasion between 16-34 weeks gestation.
  Serum insulin will be measured using commercially available assays in venous samples taken 60 min after 75g oral glucose.
  Mean serum insulin at 60 min post 75g oral glucose in pregnant women of Black (Black African and Black Caribbean) and White European ethnicity will be reported and compared using a t test.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine F Hunt, MBBS MRCP, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- Clinical Research Facility, King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No